CLINICAL TRIAL: NCT02956655
Title: Effect of Fasting Therapy on Blood Glucose Control and Islet Function in Newly Diagnosed Type 2 Diabetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jian Qin, director of the education department, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016NO.093
Record Dates: First submitted 2016-09-21; First posted 2016-11-07 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fasting therapy (Experimental): Fasting therapy, lasting for 14 days, all subjects are isolated from ordinary food. However, drinking water is not limited and they are encouraged to drink more, at least 3 liters. Besides, they need to take some middle intensity exercise for at least 2 hours. They will take some prescribed medications except for hypoglycemic drugs.
  Interventions: Other: Fasting therapy; Other: Exercise; Behavioral: Lifestyle guidance
- Insulin intensive therapy (Active Comparator): Insulin intensive therapy, receive continuous subcutaneous insulin infusion. (Human Insulin (Novolin-R, Novo Nordisk) Device: H-Tron Plus V100; Disetronic Medical System, Burgdorf, Switzerland). The insulin dose used will be adjusted everyday according to their glucose by a physician until a target blood glucose level been reached.
  Interventions: Drug: Insulin intensive therapy: Human Insulin (Novolin-R, Novo Nordisk); Other: Exercise; Behavioral: Lifestyle guidance; Device: H-Tron Plus V100; Disetronic Medical System, Burgdorf, Switzerland

INTERVENTIONS:
Other: Fasting therapy — The target fasting plasma glucose is set below 6.1mmol/l and the postprandial blood glucose below 8.0 mmol/l. After intervention, all the accomplished patients undergo a 1 year period follow-up. Lifestyle guidance will be offered throughout the follow-up.
  Arms: Fasting therapy
Drug: Insulin intensive therapy: Human Insulin (Novolin-R, Novo Nordisk) — Human Insulin (Novolin-R, Novo Nordisk)
  Device: H-Tron Plus V100; Disetronic Medical System, Burgdorf, Switzerland
  The target fasting plasma glucose is set below 6.1mmol/l and the postprandial blood glucose below 8.0 mmol/l. If the glucose target cannot be achieved within 2 weeks or the subjects are not tolerated with this therapy, these members will be exclude from the study and they will receive other treatment according the standard treatment guidelines. After intervention, all the accomplished patients will undergo a 1 year period follow-up. Lifestyle guidance will be offered throughout the follow-up.
  Arms: Insulin intensive therapy
Other: Exercise — Middle intense exercise for at least 2 hours,e.g. brisk walking or jogging
Behavioral: Lifestyle guidance — Lifestyle guidance is provided by specific physicians through phone calls
Device: H-Tron Plus V100; Disetronic Medical System, Burgdorf, Switzerland
  Arms: Insulin intensive therapy

SUMMARY:
The purpose of this study is to evaluate Effect of Fasting Therapy on Blood Glucose Control and Islet Function in Newly Diagnosed Type 2 Diabetic Patients.

DETAILED DESCRIPTION:
This study was to investigate the effects of fasting therapy on blood glucose control and islet function in newly diagnosed type 2 diabetic patients.

60 participants will be recruited from outpatients or inpatients in First Affiliated Hospital of Sun Yat-sen University according the eligibility criteria. All the eligible subjects will be randomly allocated into 2 groups, the fasting group and the intense insulin therapy group. The former one will receive fasting therapy for 14 days and the latter be treated with an intense insulin therapy including short-term continuous subcutaneous insulin infusion treatment or four stage intensive insulin treatment for 2 weeks.

First of all, to determine whether fasting therapy is effective for glucose control or not, the investigators will observed the required time and control rate for a targeted glucose level, the average fasting blood glucose and postprandial blood glucose as well as the glucose amelioration degree in all the patients. Then, all the patients will undergo a follow-up period of 1 year, during which the fasting and postprandial blood glucose and glycosylated hemoglobin of each participant will be monitored to assess the long-term remission rate of diabetes. Patients are invited to review their glucose and lipid metabolic indices at 3 months, 6 months and 12 months of follow-up. Lifestyle guidance will be offered by specialist physicians throughout the follow-up period.

Secondly, all the patients are required to take the insulin and C-peptide releasing tests before and after fasting as well as in the follow-up to investigate the short-term and long-term treatment effect of islet function through accessing the first secretion function of pancreatic island and calculating insulin resistance(HOMA-IR) and HOMA-B through homeostasis model assessment.

In summary, this study aims to explore the short-term and long-term therapeutic effects in new onset type 2 diabetes, hoping to provide a novel, effective and more convenient treatment method for them.

ELIGIBILITY:
Inclusion Criteria:

* aged from 27-65 years
* overweight or obese (body mass index[BMI] ≧25.0 kg/m2)
* The function of heart, liver, kidney is normal
* Newly diagnosed Type 2 diabetes according to the diagnostic criteria and classification of diabetes mellitus in 1999 World Health Organization standards with a fasting plasma glucose level ranged from 7.0 mmol/l to 16.7 mmol/l
* sign a consent form

Exclusion Criteria:

* Females who were pregnant or experiencing a menstrual period
* Abnormal function of heart, liver, kidney
* Aged below 25 or over 70
* Malignancy, hematopathy, active tuberculosis, peptic ulcer with gastric bleeding, binge-eating disorder, psychiatric disease, congestive heart failure, cancer or a history of cancer, unstable coronary artery disease
* With acute or severe chronic diabetic complications
* Without an informed consent
* Severe intercurrent illness
* Tested positive for glutamic acid decarboxylase antibody
* Patients with maturity onset diabetes in youth and mitochondria diabetes mellitus
* Other situations which the investigators think that it is inappropriate to include

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
The remission rate of diabetes | 6 months

SECONDARY OUTCOMES:
β-cell function--HOMA-IR | 6 months
  HOMA means "Homeostasis model assessment". It is a designed model for evaluating the extent of individual's insulin resistance. The specific calculate formula is listed as follows, "fasting plasma glucose(mmol/l) × fasting insulin(mIU/L)/22.5". So it's a specific value without measurement. The normal value of it is 1. Higher than 1 indicate insulin resistance. HOMA-B refers to the basial pancreas islet function. The formula is "20 × fasting insulin / (fasting plasma glucose-3.5)". The measurement of it is percent(%). The normal value of it is 100%. The value of it will decrease when the patients's pancreas islet function is worse.
β-cell function--HOMA-B (%) | 6 months
  HOMA means "Homeostasis model assessment". It is a designed model for evaluating the extent of individual's insulin resistance. The specific calculate formula is listed as follows, "fasting plasma glucose(mmol/l) × fasting insulin(mIU/L)/22.5". So it's a specific value without measurement. The normal value of it is 1. Higher than 1 indicate insulin resistance. HOMA-B refers to the basial pancreas islet function. The formula is "20 × fasting insulin / (fasting plasma glucose-3.5)". The measurement of it is percent(%). The normal value of it is 100%. The value of it will decrease when the patients's pancreas islet function is worse.
Weight (kg) | before enrollment, after the intervention (at day 14th), 6 month after the intervention
BMI (kg/m^2) | before enrollment, after the intervention (at day 14th), 6 month after the intervention
Lipid profile (mmol/l) | before enrollment, after the intervention (at day 14th), 6 month after the intervention
Uric acid (mmol/l) | before enrollment, after the intervention (at day 14th), 6 month after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jian Qin, Doctor, Study Director — Sun Yat-sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No